CLINICAL TRIAL: NCT00435409
Title: A Randomized, Phase 3 Study Of Sunitinib In Combination With Capecitabine Compared With Capecitabine In Patients With Previously Treated Breast Cancer
Brief Title: A Study Of Sunitinib In Combination With Capecitabine Compared With Capecitabine In Patients With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A6181099
Record Dates: First submitted 2007-02-13; First posted 2007-02-15 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Sunitinib + Capecitabine
- B (Active Comparator)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Sunitinib + Capecitabine — Sunitinib administered orally at a starting dose of 37.5 mg once a day on a continuous regimen.
  Capecitabine administered orally at a starting dose of 2000 mg/m^2 per day [1000 mg/m^2 bid (twice daily)] from days 1-14 every 3 weeks. Study treatment should be given until progression or withdrawal from the study for other reasons.
  Arms: A
Drug: Capecitabine — Capecitabine administered orally at a starting dose of 2500 mg/m^2 per day [1250 mg/m^2 bid (twice daily)] from days 1-14 every 3 weeks. Study treatment should be given until progression or withdrawal from the study for other reasons. At the time of progression, patients may be eligible to crossover to single agent sunitinib, administered orally at a starting dose of 37.5 mg daily.
  Arms: B

SUMMARY:
The treatment received with sunitinib plus capecitabine could delay tumor growth longer than with treatment with capecitabine alone.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic disease that can be measured. Patients with bone-only disease are also allowed to enter the study.
* Previous treatment with an anthracycline and a taxane in any setting
* Progression on first or second line regimen or adjuvant regimen if disease free interval less than 12 months

Exclusion Criteria:

* History of inflammatory carcinoma if there is no other measurable disease
* More than 2 chemotherapy agents in the advanced disease setting
* Brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (136):
- United States (59):
  - Pfizer Investigational Site, Downey, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Montebello, California
  - Pfizer Investigational Site, Whittier, California
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Boynton Beach, Florida
  - Pfizer Investigational Site, Coral Springs, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Lakeland, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Duluth, Georgia
  - Pfizer Investigational Site, Lawrenceville, Georgia
  - Pfizer Investigational Site, Snellville, Georgia
  - Pfizer Investigational Site, Avon, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Mooresville, Indiana
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Gretna, Louisiana
  - Pfizer Investigational Site, Marrero, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Kensington, Maryland
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Clairton, Pennsylvania
  - Pfizer Investigational Site, Greensburg, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Pottstown, Pennsylvania
  - Pfizer Investigational Site, Wexford, Pennsylvania
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Gallatin, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Smyrna, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Georgetown, Texas
  - Pfizer Investigational Site, Bountiful, Utah
  - Pfizer Investigational Site, Layton, Utah
  - Pfizer Investigational Site, Murray, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Provo, Utah
  - Pfizer Investigational Site, West Valley City, Utah
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Kennewick, Washington
- Austria (3):
  - Pfizer Investigational Site, Linz
  - Pfizer Investigational Site, Salzburg
  - Pfizer Investigational Site, Wels
- Belgium (5):
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Namur
  - Pfizer Investigational Site, Turnhout
  - Pfizer Investigational Site, Yvoir
- Canada (3):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Pfizer Investigational Site, Prague, Czechia
- Denmark (3):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Koebenhavn OE
  - Pfizer Investigational Site, Odense
- France (7):
  - Pfizer Investigational Site, Montpellier, Cedex 05
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Paris
- Germany (10):
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Frankenthal
  - Pfizer Investigational Site, Frankfurt am Main
  - Pfizer Investigational Site, Fürstenwalde
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Nuremberg
  - Pfizer Investigational Site, Stendal
  - Pfizer Investigational Site, Ulm
  - Pfizer Investigational Site, Völklingen
- Greece (5):
  - Pfizer Investigational Site, Heraklion, Crete
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Ioannina
  - Pfizer Investigational Site, Pátrai
  - Pfizer Investigational Site, Thessaloniki
- Pfizer Investigational Site, Dublin, Ireland
- Italy (9):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Messina
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Saronno (VA)
  - Pfizer Investigational Site, Torino
- Netherlands (3):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Sittard-geleen
  - Pfizer Investigational Site, Zwolle
- Norway (2):
  - Pfizer Investigational Site, Levanger
  - Pfizer Investigational Site, Oslo
- Poland (3):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Warsaw
- Romania (2):
  - Pfizer Investigational Site, Cluj-Napoca, Cluj
  - Pfizer Investigational Site, Bucharest, Sector 2
- Russia (3):
  - Pfizer Investigational Site, Kuzmolovo, Vsevolozhsk District, Leningradskaya Oblast'
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Spain (6):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Burgos, Burgos
  - Pfizer Investigational Site, Cadiz, Cadiz
  - Pfizer Investigational Site, A Coruña, La Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla
- United Kingdom (11):
  - Pfizer Investigational Site, Truro, Cornwall
  - Pfizer Investigational Site, Chelmsford, Essex
  - Pfizer Investigational Site, Harlow, Essex
  - Pfizer Investigational Site, Burton-on-Trent, Staffordshire
  - Pfizer Investigational Site, Worthing, West Sussex
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Essex
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Swansea
  - Pfizer Investigational Site, Truro
  - Pfizer Investigational Site, Worthing

REFERENCES:
- [Derived] Crown JP, Dieras V, Staroslawska E, Yardley DA, Bachelot T, Davidson N, Wildiers H, Fasching PA, Capitain O, Ramos M, Greil R, Cognetti F, Fountzilas G, Blasinska-Morawiec M, Liedtke C, Kreienberg R, Miller WH Jr, Tassell V, Huang X, Paolini J, Kern KA, Romieu G. Phase III trial of sunitinib in combination with capecitabine versus capecitabine monotherapy for the treatment of patients with pretreated metastatic breast cancer. J Clin Oncol. 2013 Aug 10;31(23):2870-8. doi: 10.1200/JCO.2012.43.3391. Epub 2013 Jul 15. PMID 23857972
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181099&StudyName=A%20Study%20Of%20Sunitinib%20In%20Combination%20With%20Capecitabine%20Compared%20With%20Capecitabine%20In%20Patients%20With%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib + Capecitabine: Sunitinib administered orally at a starting dose of 37.5 milligrams (mg) once a day on a continuous regimen. Capecitabine administered orally at a starting dose of 2000 milligrams per square meter (mg/m^2) per day (1000 mg/m^2 twice daily [BID]) from Days 1-14 every 3 weeks.
- Capecitabine, no Crossover: Capecitabine administered orally at a starting dose of 2500 mg/m^2 per day (1250 mg/m^2 BID) from Days 1-14 every 3 weeks.
- Capecitabine, Crossover to Sunitinib: Capecitabine administered orally at a starting dose of 2500 mg/m^2 per day (1250 mg/m^2 BID) from Days 1-14 every 3 weeks. At the time of progression, crossover to single agent sunitinib, administered orally at a starting dose of 37.5 mg daily continuously.
Period: Overall Study
Arm/Group | Sunitinib + Capecitabine | Capecitabine, no Crossover | Capecitabine, Crossover to Sunitinib
Started | 221 | 143 | 78
Treated | 217 | 139 | 78
Completed | 0 | 0 | 0
Not Completed | 221 | 143 | 78
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Death | 8 | 6 | 6
Not completed — Objective progression or relapse | 158 | 93 | 58
Not completed — Global deterioration of health status | 0 | 0 | 4
Not completed — Withdrawal by Subject | 8 | 7 | 1
Not completed — Other | 45 | 30 | 1
Not completed — Adverse Event | 0 | 0 | 8
Not completed — Sponsor decision | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib + Capecitabine: Sunitinib administered orally at a starting dose of 37.5 mg once a day on a continuous regimen. Capecitabine administered orally at a starting dose of 2000 mg/m^2 per day (1000 mg/m^2 BID) from Days 1-14 every 3 weeks.
- Capecitabine: Capecitabine administered orally at a starting dose of 2500 mg/m^2 per day (1250 mg/m^2 BID) from Days 1-14 every 3 weeks. At the time of progression, participants could have been eligible to crossover to single agent sunitinib, administered orally at a starting dose of 37.5 mg daily continuously.
- Total: Total of all reporting groups
Arm/Group | Sunitinib + Capecitabine | Capecitabine | Total
Number analyzed (Participants) | 221 | 221 | 442
Age, Customized [Number; unit: participants]
  Less than 65 years | 182 | 185 | 367
  Greater than or equal to 65 years | 39 | 36 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 220 | 438
  Male | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Defined as the time from the date of randomization to the date of the first documentation of objective tumor progression or death due to any cause, whichever occurs first. If tumor progression data include more than 1 date, the first date will be used. PFS (in months) will be calculated as (first event date minus randomization date plus 1) divided by 30.4.
Time Frame: Baseline until disease progression (up to 3 years from first dose)
Population: Intent to treat (ITT) population: defined as all participants who were randomized
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib + Capecitabine | Capecitabine
Number analyzed (Participants) | 221 | 221
months
  Independent radiology assessment | 5.5 [4.5 to 6.0] | 5.9 [5.4 to 7.6]
  Investigator's assessment | 5.4 [4.4 to 5.8] | 5.5 [4.3 to 6.8]
Statistical Analysis 1: Comparison: Sunitinib + Capecitabine vs Capecitabine; A stratified log-rank test (1-sided, α=0.025) based on randomization stratification factors; Test type: Superiority or Other; p = 0.9409, Log Rank — Stratification factors included metastatic organ sites (2 or less versus [vs] more than [>] 2 sites), hormone receptor status (HER2-/ER-/PR-) vs all others), and prior chemotherapy regimens (1 vs >1), from interactive voice response system (IVRS); Hazard Ratio (HR) = 1.2239, 95% CI 2-sided [0.9487 to 1.5789]
Statistical Analysis 2: Comparison: Sunitinib + Capecitabine vs Capecitabine; A stratified log-rank test (1-sided, α=0.025) based on randomization stratification factors; Test type: Superiority or Other; p = 0.8120, Log Rank — Stratification factors include metastatic organ sites (2 or less versus [vs] 2 or more sites), hormone receptor status (HER2-/ER-/PR-) vs all others), and prior chemotherapy regimens (1 vs more than 1), from IVRS; Hazard Ratio (HR) = 1.1084, 95% CI 2-sided [0.8817 to 1.3935]

2. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Proportion of participants with confirmed complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST); CR: disappearance of all target lesions, PR: greater than or equal to (>=) 30 percent (%) decrease in the sum of the longest dimensions (SLD) of the target lesions taking as a reference the baseline SLD. Confirmed responses = persist on repeat imaging study at least 4 weeks after initial documentation of response. Designation of best response of stable disease (SD) required the criteria to be met at least 5 weeks after randomization.
Time Frame: Baseline until response or disease progression (up to 3 years from first dose)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib + Capecitabine | Capecitabine
Number analyzed (Participants) | 221 | 221
percentage of participants
  Independent radiology assessment | 18.6 [13.7 to 24.3] | 16.3 [11.7 to 21.8]
  Investigator's assessment | 25.3 [19.7 to 31.6] | 20.4 [15.3 to 26.3]
Statistical Analysis 1: Comparison: Sunitinib + Capecitabine vs Capecitabine; Independent radiology assessment; Test type: Superiority or Other; p = 0.3143, Cochran-Mantel-Haenszel — A stratified CMH test stratified by randomization stratification factors was used to compare objective response rate (ORR) between two treatment arms; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.69 to 1.97]
Statistical Analysis 2: Comparison: Sunitinib + Capecitabine vs Capecitabine; Investigator's assessment; Test type: Superiority or Other; p = 0.1269, Cochran-Mantel-Haenszel — A stratified CMH test stratified by randomization stratification factors was used to compare ORR between two treatment arms; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.83 to 2.13]

3. Secondary Outcome: Duration of Response (DR)
Description: Time from the first documentation of objective tumor response (CR or PR) that was subsequently confirmed to the first documentation of disease progression (PD) or to death due to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. DR (in months) was calculated as [the date response ended (date of PD or death) minus first CR or PR date that was subsequently confirmed plus 1)] divided by 30.4.
Time Frame: Baseline until response or disease progression (up to 3 years from first dose)
Population: ITT subgroup of participants with a confirmed objective tumor response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib + Capecitabine | Capecitabine
Number analyzed (Participants) | 41 | 36
months
  Independent radiology assessment | 9.0 [5.7 to 20.7] | 8.8 [5.7 to 13.8]
  Investigator's assessment | 5.7 [4.3 to 6.9] | 7.6 [6.5 to 9.9]

4. Secondary Outcome: Overall Survival (OS)
Description: Time from the date of randomization to the date of death due to any cause. OS (in months) calculated as (date of death minus randomization date plus 1) divided by 30.4. For patients lacking survival data beyond the date of their last follow-up, the OS time was censored on the last date they were known to be alive. Patients lacking survival data beyond randomization had their OS times censored at randomization.
Time Frame: Baseline until death or up to 3 years from first dose
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib + Capecitabine | Capecitabine
Number analyzed (Participants) | 221 | 221
months | 16.5 [14.5 to 19.6] | 17.2 [15.5 to 19.3]
Statistical Analysis 1: Comparison: Sunitinib + Capecitabine vs Capecitabine; Test type: Superiority or Other; p = 0.6275, Log Rank — Stratification factors (all from IVRS) included number of metastatic organ sites (<=2 vs >2 sites), hormone receptor status (HER2-/ER-/PR- vs all others), and prior chemotherapy regimens (1 vs >1); Hazard Ratio (HR) = 1.0372, 95% CI 2-sided [0.8322 to 1.2927] — Hazard ratio for sunitinib + capecitabine versus capecitabine

5. Secondary Outcome: Percent Chance of Participant Survival
Description: Probability of survival 2 years and 3 years after the first dose of study treatment.
Time Frame: Year 1, Year 2, Year 3
Population: ITT population
Measure: Number (95% Confidence Interval); unit: probability of survival
Arm/Group | Sunitinib + Capecitabine | Capecitabine
Number analyzed (Participants) | 221 | 221
probability of survival
  Year 1 | 0.635 [0.567 to 0.696] | 0.654 [0.585 to 0.715]
  Year 2 | 0.368 [0.303 to 0.433] | 0.373 [0.306 to 0.440]
  Year 3 | 0.150 [0.098 to 0.213] | 0.174 [0.115 to 0.243]

6. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer's Quality of Life Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30: global health/quality of life (QoL), functional domains (physical, role, cognitive, emotional, social), and symptom scales/items (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea). Recall period: past week; response range: not at all to very much; global/QoL range: very poor to excellent. Scale score range: 0 to 100. Higher functional/global QoL score = better functioning and higher symptom score = greater degree of symptoms
Time Frame: Day 1 of each treatment cycle (up to 3 years or end of treatment)
Population: Patient Reported Outcomes (PRO) assessments were not analyzed because the study did not meet its primary endpoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sunitinib + Capecitabine | Capecitabine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer's Quality of Life Questionnaire Breast Cancer Module (EORTC QLQ-BR23)
Description: BR23: measured disease related symptoms of dry mouth, eye pain, hair loss, hot flushes, attractiveness, future health, sexual activity, arm/shoulder pain, breast pain, swollen breast, and skin problems on the breast. Recall period: past week; response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
Time Frame: Day 1 of each treatment cycle (up to 3 years or end of treatment)
Population: PRO assessments were not analyzed because the study did not meet its primary endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sunitinib + Capecitabine | Capecitabine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in EuroQol Group's EuroQol 5-Dimensional Self-Report Questionnaire (EQ-5D)
Description: EQ-5D: health status in 5 dimensions (mobility, self-care, pain/discomfort, anxiety/depression, usual activities). Three-level scale (1=no problem, 2=some problem, and 3=extreme problem). A single score between 1 and 3 is generated for each domain. For each subject, the outcome rating on the 5 domains could be mapped to a single index through an algorithm. The index ranges between 0 and 1, with the higher score indicating a better health state perceived by the participant.
Time Frame: Day 1 of each treatment cycle (up to 3 years or end of treatment)
Population: PRO assessments were not analyzed because the study did not meet its primary endpoint.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Sunitinib + Capecitabine | Capecitabine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib + Capecitabine | Capecitabine
Serious Adverse Events (participants affected / at risk) | 85/217 | 59/215
Other Adverse Events (participants affected / at risk) | 214/217 | 208/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Capecitabine (N=217) | Capecitabine (N=215)
Anaemia (Blood and lymphatic system disorders) | 7 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 9 | 13
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 1
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 6
Asthenia (General disorders) | 6 | 0
Chest pain (General disorders) | 1 | 2
Chills (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 10 | 7
Fatigue (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 3 | 1
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 6
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Breast infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 3
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram ST segment depression (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 1 | 0
Diabetic coma (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal infarct (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 3
Ureteral catheterisation (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Iliac artery thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Ulcer (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
HAEMATEMESIS SECONDARY TO THROMBCYTOPENIA (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Capecitabine (N=217) | Capecitabine (N=215)
Anaemia (Blood and lymphatic system disorders) | 53 | 35
Leukopenia (Blood and lymphatic system disorders) | 51 | 19
Neutropenia (Blood and lymphatic system disorders) | 104 | 39
Thrombocytopenia (Blood and lymphatic system disorders) | 102 | 14
Hypothyroidism (Endocrine disorders) | 22 | 2
Conjunctivitis (Eye disorders) | 4 | 16
Lacrimation increased (Eye disorders) | 23 | 24
Abdominal pain (Gastrointestinal disorders) | 38 | 29
Abdominal pain upper (Gastrointestinal disorders) | 48 | 30
Constipation (Gastrointestinal disorders) | 41 | 42
Diarrhoea (Gastrointestinal disorders) | 121 | 95
Dry mouth (Gastrointestinal disorders) | 19 | 16
Dyspepsia (Gastrointestinal disorders) | 38 | 13
Dysphagia (Gastrointestinal disorders) | 13 | 1
Flatulence (Gastrointestinal disorders) | 13 | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 | 5
Gingivitis (Gastrointestinal disorders) | 11 | 2
Nausea (Gastrointestinal disorders) | 122 | 91
Oesophagitis (Gastrointestinal disorders) | 14 | 2
Stomatitis (Gastrointestinal disorders) | 61 | 26
Vomiting (Gastrointestinal disorders) | 90 | 55
Asthenia (General disorders) | 75 | 49
Chest pain (General disorders) | 12 | 12
Fatigue (General disorders) | 65 | 53
Mucosal inflammation (General disorders) | 49 | 24
Oedema peripheral (General disorders) | 16 | 19
Pain (General disorders) | 11 | 8
Pyrexia (General disorders) | 21 | 15
Hyperbilirubinaemia (Hepatobiliary disorders) | 13 | 13
Jaundice (Hepatobiliary disorders) | 11 | 0
Nasopharyngitis (Infections and infestations) | 16 | 10
Rhinitis (Infections and infestations) | 1 | 13
Urinary tract infection (Infections and infestations) | 16 | 11
Alanine aminotransferase increased (Investigations) | 11 | 15
Aspartate aminotransferase increased (Investigations) | 19 | 13
Blood alkaline phosphatase increased (Investigations) | 12 | 8
Platelet count decreased (Investigations) | 15 | 4
Weight decreased (Investigations) | 20 | 17
Decreased appetite (Metabolism and nutrition disorders) | 67 | 44
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 25
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 23
Bone pain (Musculoskeletal and connective tissue disorders) | 13 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 33
Dizziness (Nervous system disorders) | 14 | 9
Dysgeusia (Nervous system disorders) | 58 | 18
Headache (Nervous system disorders) | 57 | 32
Neuropathy peripheral (Nervous system disorders) | 9 | 13
Paraesthesia (Nervous system disorders) | 15 | 16
Peripheral sensory neuropathy (Nervous system disorders) | 16 | 6
Anxiety (Psychiatric disorders) | 14 | 10
Insomnia (Psychiatric disorders) | 18 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 28
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 31 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 16
Erythema (Skin and subcutaneous tissue disorders) | 15 | 12
Nail disorder (Skin and subcutaneous tissue disorders) | 14 | 19
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 118 | 131
Rash (Skin and subcutaneous tissue disorders) | 18 | 24
Skin fissures (Skin and subcutaneous tissue disorders) | 3 | 12
Hot flush (Vascular disorders) | 11 | 6
Hypertension (Vascular disorders) | 46 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 2 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 5 | 0
Macrocytosis (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 3 | 0
Arrhythmia (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 4 | 1
Palpitations (Cardiac disorders) | 4 | 1
Pericardial effusion (Cardiac disorders) | 3 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 4
Tachycardia (Cardiac disorders) | 2 | 2
Ear pain (Ear and labyrinth disorders) | 4 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 3
Vertigo (Ear and labyrinth disorders) | 8 | 13
Hyperthyroidism (Endocrine disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Conjunctival irritation (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 2 | 0
Dry eye (Eye disorders) | 7 | 4
Exophthalmos (Eye disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 0
Eye inflammation (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 5 | 7
Eye oedema (Eye disorders) | 2 | 2
Eye pain (Eye disorders) | 2 | 1
Eye swelling (Eye disorders) | 1 | 0
Eyelash discolouration (Eye disorders) | 2 | 0
Eyelid oedema (Eye disorders) | 5 | 0
Eyelid ptosis (Eye disorders) | 1 | 1
Keratitis (Eye disorders) | 1 | 0
Mydriasis (Eye disorders) | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Ocular icterus (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 2 | 0
Photophobia (Eye disorders) | 0 | 1
Retinal disorder (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 2
Visual acuity reduced (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 9 | 1
Vitreous floaters (Eye disorders) | 2 | 0
Xerophthalmia (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Eye disorders) | 2 | 4
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 1 | 2
Anal inflammation (Gastrointestinal disorders) | 4 | 0
Anal stenosis (Gastrointestinal disorders) | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 8 | 5
Ascites (Gastrointestinal disorders) | 5 | 2
Chapped lips (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 3
Colitis (Gastrointestinal disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Eructation (Gastrointestinal disorders) | 4 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 9 | 1
Gingival disorder (Gastrointestinal disorders) | 1 | 0
Gingival oedema (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 4 | 1
Gingival swelling (Gastrointestinal disorders) | 1 | 0
Gingival ulceration (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 2 | 0
Glossodynia (Gastrointestinal disorders) | 6 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 5 | 7
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 3
Lip haematoma (Gastrointestinal disorders) | 0 | 1
Lip pain (Gastrointestinal disorders) | 1 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 4 | 1
Odynophagia (Gastrointestinal disorders) | 2 | 0
Oedema mouth (Gastrointestinal disorders) | 1 | 0
Oesophageal disorder (Gastrointestinal disorders) | 1 | 1
Oesophageal pain (Gastrointestinal disorders) | 1 | 2
Oral discomfort (Gastrointestinal disorders) | 3 | 0
Oral mucosal eruption (Gastrointestinal disorders) | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 8 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 7 | 2
Reflux oesophagitis (Gastrointestinal disorders) | 2 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 2 | 2
Tongue discolouration (Gastrointestinal disorders) | 1 | 1
Tongue oedema (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 5 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Axillary pain (General disorders) | 8 | 3
Catheter site pain (General disorders) | 0 | 1
Catheter site rash (General disorders) | 1 | 0
Chest discomfort (General disorders) | 2 | 1
Chills (General disorders) | 5 | 3
Condition aggravated (General disorders) | 1 | 2
Disease progression (General disorders) | 1 | 0
Face oedema (General disorders) | 6 | 2
Feeling abnormal (General disorders) | 1 | 0
Feeling cold (General disorders) | 2 | 1
Feeling hot (General disorders) | 1 | 0
Gait disturbance (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 3 | 3
Hyperthermia (General disorders) | 3 | 0
Induration (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Influenza like illness (General disorders) | 3 | 6
Infusion site extravasation (General disorders) | 0 | 1
Injection site thrombosis (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Localised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Mass (General disorders) | 0 | 1
Nodule (General disorders) | 1 | 1
Oedema (General disorders) | 4 | 2
Secretion discharge (General disorders) | 1 | 0
Swelling (General disorders) | 0 | 1
Temperature intolerance (General disorders) | 1 | 0
Thirst (General disorders) | 0 | 1
Ulcer (General disorders) | 1 | 2
Xerosis (General disorders) | 3 | 3
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 2 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 2
Abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 7 | 7
Bronchopneumonia (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 3
Clostridial infection (Infections and infestations) | 1 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 5 | 6
Device related infection (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 0 | 2
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 5
Herpes simplex (Infections and infestations) | 4 | 3
Herpes virus infection (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 7 | 7
Laryngitis (Infections and infestations) | 3 | 3
Localised infection (Infections and infestations) | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 4
Lung infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 1
Nail bed infection (Infections and infestations) | 1 | 2
Nail infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 2 | 0
Onychomycosis (Infections and infestations) | 0 | 2
Oral candidiasis (Infections and infestations) | 1 | 3
Oral fungal infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 3
Oral infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Otitis media (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 4 | 5
Puncture site infection (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 3
Skin infection (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 3
Tooth abscess (Infections and infestations) | 9 | 4
Tooth infection (Infections and infestations) | 4 | 0
Tracheitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Vaginal infection (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 1 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 3 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 1
Vulvovaginitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 2
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Whiplash injury (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 6 | 3
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood iron increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood phosphorus decreased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 2 | 2
Blood pressure decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 7 | 4
Blood uric acid increased (Investigations) | 2 | 1
Breath sounds abnormal (Investigations) | 0 | 2
Creatinine renal clearance decreased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 8 | 3
Electrocardiogram QT prolonged (Investigations) | 2 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 1
Haemoglobin (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 2
Heart rate increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 1
Protein total increased (Investigations) | 0 | 1
Respiratory rate increased (Investigations) | 0 | 1
Thyroid function test abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 1
Weight increased (Investigations) | 2 | 5
White blood cell count decreased (Investigations) | 7 | 2
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1
Tetany (Metabolism and nutrition disorders) | 1 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 4 | 3
Joint lock (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 10 | 10
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 2
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 2
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance disorder (Nervous system disorders) | 2 | 0
Burning sensation (Nervous system disorders) | 2 | 0
Cervical root pain (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0
Dysaesthesia (Nervous system disorders) | 8 | 8
Formication (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 2 | 0
Hypersomnia (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 4 | 6
Hypogeusia (Nervous system disorders) | 1 | 0
Hypokinesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 4
Migraine (Nervous system disorders) | 4 | 2
Neuralgia (Nervous system disorders) | 1 | 2
Neurotoxicity (Nervous system disorders) | 1 | 0
Paresis (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 3 | 2
Polyneuropathy (Nervous system disorders) | 3 | 3
Presyncope (Nervous system disorders) | 1 | 1
Radicular syndrome (Nervous system disorders) | 1 | 0
Radiculitis lumbosacral (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 4
Sensory disturbance (Nervous system disorders) | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 9 | 2
Speech disorder (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 2
Trigeminal nerve disorder (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 1
Apathy (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 4 | 2
Delirium (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 4 | 4
Disorientation (Psychiatric disorders) | 1 | 0
Emotional disorder (Psychiatric disorders) | 0 | 1
Emotional distress (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 2 | 0
Nervousness (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 2
Stress (Psychiatric disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 2 | 2
Chromaturia (Renal and urinary disorders) | 4 | 0
Dysuria (Renal and urinary disorders) | 6 | 3
Haematuria (Renal and urinary disorders) | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Renal pain (Renal and urinary disorders) | 1 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1
Breast discharge (Reproductive system and breast disorders) | 1 | 0
Breast induration (Reproductive system and breast disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Breast oedema (Reproductive system and breast disorders) | 2 | 0
Breast pain (Reproductive system and breast disorders) | 8 | 8
Breast swelling (Reproductive system and breast disorders) | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 5 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 2
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Retracted nipple (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 9 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 | 1
Hyperkeratosis palmaris and plantaris (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 1
Madarosis (Skin and subcutaneous tissue disorders) | 2 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 3
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 7
Purpura (Skin and subcutaneous tissue disorders) | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 0 | 1
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 7 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 6 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 3
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 2
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 9 | 0
Inadequate diet (Social circumstances) | 1 | 0
Breast reconstruction (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 1
Capillary fragility (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 4
Flushing (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 6 | 0
Hyperaemia (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 9
Intermittent claudication (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 3 | 10
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 3
Phlebitis (Vascular disorders) | 1 | 2
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 0
Trousseau's syndrome (Vascular disorders) | 1 | 1
Vasoconstriction (Vascular disorders) | 1 | 0
Venous insufficiency (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.